CLINICAL TRIAL: NCT06686771
Title: Consolidative Use of Radiotherapy to Block (CURB2) Oligoprogression In Patients With Metastatic Non-Small-Cell Lung Cancer
Brief Title: Radiotherapy to Block Oligoprogression In Metastatic Non-Small-Cell Lung Cancer
Acronym: CURB2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: Alliance for Clinical Trials in Oncology (Other); ECOG-ACRIN Cancer Research Group (Network); NRG Oncology (Other); SWOG Cancer Research Network (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCTG-BR38; CCTG-BR38 (Other: NCI CTRP); NCI-2024-09093 (Other: NCI/CTEP)
Record Dates: First submitted 2024-11-11; First posted 2024-11-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- SBRT/Radiotherapy followed by standard of care therapy (Experimental)
  Interventions: Radiation: SBRT
- No SBRT and switch to second-line standard of care therapy (Active Comparator)
  Interventions: Other: Second-line standard of care therapy

INTERVENTIONS:
Radiation: SBRT — Please refer to the current NCCN NSCLC guidelines for possible treatment options
  Arms: SBRT/Radiotherapy followed by standard of care therapy
Other: Second-line standard of care therapy — Please refer to the current NCCN NSCLC guidelines for possible treatment options.
  Arms: No SBRT and switch to second-line standard of care therapy

SUMMARY:
This study is being done to answer the following question: Can the chance of lung cancer growing or spreading be lowered by adding targeted radiotherapy to the usual combination of drugs?

This study is being done to find out if this approach is better or worse than the usual approach for lung cancer. The usual approach is defined as the care most people get for non-small cell lung cancer.

DETAILED DESCRIPTION:
The usual approach for patients who are not in a study and whose disease has gotten worse is to switch treatments. Sometimes, combinations of drugs or radiotherapy are used. The study doctor can explain which treatment may be best. These treatments can reduce symptoms and may stop the tumour from growing for several months or longer.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic disease (stage IV) detected on imaging and histologically and/or cytologically confirmed NSCLC as per the WHO Classification of Tumors and AJCC 8th Edition TNM Classification, without an actionable driver mutation, for whom either ICI alone or combination ICI + chemotherapy is indicated
* Oligoprogression on first-line ICI +/- chemotherapy systemic therapy after at least 3 cycles.
* All sites of oligoprogression can be safely treated with SBRT or ablative radiotherapy as determined by radiation treatment preplan, including availability and tolerability of necessary technologies (e.g., active breathing control, MRLinac, fiducial insertion, etc.) and accounting for previous radiotherapy overlap. Safety must be assessed and determined by a radiation oncologist.
* Patients with treated CNS disease who have radiologic and clinical evidence of stable brain metastases, with no evidence of cavitation or hemorrhage in the brain lesion, are eligible providing that they are asymptomatic and do not require corticosteroids (must have discontinued steroids at least 1 week prior to randomization).
* Candidate for regulatory approved SOC second-line systemic therapy options if randomized to Arm 2.
* Participants must be ≥ 18 years of age.
* ECOG performance status of 0, 1 or 2.
* Participants that received prior adjuvant/neoadjuvant/consolidation systemic therapy (including chemotherapy and ICI ) are eligible if at least 6 months have elapsed between the completion of prior therapy and start of first-line treatment for metastatic disease.
* Participants must have recovered to ≤ grade 1 from all reversible toxicity related to prior systemic therapy.
* Previous surgery related to NSCLC in the curative or metastatic disease setting is permitted. Previous major surgery is permitted provided that surgery occurred at least 28 days prior to participant enrollment and that wound healing has occurred.
* Prior external beam radiation related to NSCLC in the metastatic disease setting is permitted provided a minimum of 14 days (2 weeks) have elapsed between the last dose of radiation and date of enrollment. Patients that received prior external beam radiation therapy in the NSCLC curative disease setting (including the primary lesion) are eligible. Oligoprogressive lesions previously treated with external beam radiation are eligible as long they are clinically asymptomatic, and re-treatment is possible according to the investigator.
* Prior conventional, non-stereotactic radiotherapy for palliative purposes is allowed, and if the palliated lesion subsequently progressed but asymptomatic not requiring immediate RT, the lesion can still be counted toward one of the five oligoprogressive lesions.
* For Arm 1, SBRT must be initiated within 3 weeks of participant enrollment.
* Participant is able (i.e. sufficiently fluent) and willing to complete the quality of life and/or health utility questionnaires in either English, French, or Spanish.
* Reimbursement of continued SOC ICI and chemotherapy systemic therapies may not be uniform across all sites. In the event that site/investigator is unable to provide access to the drug, participant will not be eligible for this trial.
* Participants must be accessible for treatment and follow-up. Investigators must assure themselves the participants enrolled on this trial will be available for complete documentation of the treatment, adverse events, and follow-up.
* Participants of childbearing potential must have agreed to use a highly effective contraceptive method.

Exclusion Criteria:

* Large-cell neuroendocrine carcinoma (LCNEC), pulmonary carcinoid tumour or mixed small cell and non-small cell lung cancer are not eligible.
* Presence of leptomeningeal disease.
* Pregnancy.
* Serious medical conditions in which radiotherapy of target lesions is contraindicated (e.g., scleroderma, Ataxia Telangiectasia (ATM), interstitial lung disease (ILD), Child-Pugh C liver function).
* Any other condition in which in the judgement of the investigator would make the patient inappropriate for study entry.
* Patients who are not on actively on ICI or ICI + chemotherapy.
* Participants with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Concomitant medications should only exclude participants from trial participation when clinically relevant known or predicted drug-drug interactions or potential overlapping toxicities will impact safety or efficacy; please consult the relevant product monographies.
* Concurrent treatment with other anti-cancer therapy, including investigational agents.
* Live attenuated vaccination administered within 30 days prior to enrollment/randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2025-12-16 (Actual); Primary Completion 2030-02-28 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 5.5 years
Overall survival | 5.5 years

SECONDARY OUTCOMES:
Number and severity of adverse events | 5.5 years
Patient-reported adverse events utilizing PRO-CTCAE questionnaire | 5.5 years
Patient-reported quality of life utilizing EORTC-QLQ-C30 questionnaire | 5.5 years
Patient-reported quality of life utilizing QLQ-LC-13 questionnaire | 5.5 years
Cost-effectiveness utilizing EQ-5D-5L questionnaire (Canadian sites only) | 5.5 years

CONTACTS AND LOCATIONS:
Overall Officials: C. Jillian Tsai, Study Chair — University Health Network Princess Margaret Hospital, Toronto, ON Canada
Locations (49):
- United States (47):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - City of Hope at Irvine Lennar, Irvine, California
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Alton Memorial Hospital, Alton, Illinois
  - Northwestern University, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - Northwestern Medicine Glenview Outpatient Center, Glenview, Illinois
  - Northwestern Medicine Grayslake Outpatient Center, Grayslake, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - HSHS Saint Elizabeth's Hospital, O'Fallon, Illinois
  - Northwestern Medicine Oak Brook, Oak Brook, Illinois
  - Northwestern Medicine Orland Park, Orland Park, Illinois
  - Memorial Hospital East, Shiloh, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Mercy Hospital, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Nebraska Medicine-Bellevue, Bellevue, Nebraska
  - Nebraska Medicine-Village Pointe, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Mount Sinai Chelsea, New York, New York
  - Mount Sinai West, New York, New York
  - Mount Sinai Hospital, New York, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Geisinger Medical Oncology-Lewisburg, Lewisburg, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Geisinger Wyoming Valley/Henry Cancer Center, Wilkes-Barre, Pennsylvania
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Northwest Wisconsin Cancer Center, Ashland, Wisconsin
- Canada (2):
  - Odette Cancer Centre- Sunnybrook Health Sciences Centre, Toronto, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: Yes
Individual patient data may be shared once the final analysis is complete following the Canadian Cancer Trials Group Data Sharing Policy
URL: https://www.ctg.queensu.ca/docs/public/policies/DataSharingandAccessPolicy.pdf